CLINICAL TRIAL: NCT01162720
Title: Feasibility of Tourniquet Use During Cement Fixation Only for TKR Surgery
Brief Title: Short- Versus Long-duration Tourniquet Use During Total Knee Replacement (TKR)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The risk of donor blood transfusion was unacceptably high in the Short Duration Group
Sponsor: Fairfield Hospital, Australia (Other)
Responsible Party: Dr Jay Dave, Fairfield Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FairfieldHJCD; 2008-15 (Other: SSWAHS)
Record Dates: First submitted 2010-07-06; First posted 2010-07-15 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Primary knee replacement; Unilateral knee replacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short duration tourniquet (Experimental): Patients allocated to this group will have the pneumatic tourniquet applied to the index limb for approximately 20-30 minutes during cement fixation of the prosthesis.
  Interventions: Procedure: Short duration tourniquet
- Long duration tourniquet (Active Comparator): Patients randomised to this arm will have the tourniquet applied from commencement of surgery and removed just prior to skin closure.
  Interventions: Procedure: Long duration tourniquet

INTERVENTIONS:
Procedure: Long duration tourniquet — Patients randomised to this arm will have the tourniquet applied at the commencement of surgery and removed prior to wound closure.
  Arms: Long duration tourniquet
Procedure: Short duration tourniquet — Patients assigned to this arm will have the tourniquet applied during cement fixation of the prosthesis only (ie removed just prior to wound closure).
  Arms: Short duration tourniquet

SUMMARY:
To establish whether a short duration of tourniquet application (from cement fixation to cement setting)is associated with better patient functional outcomes compared to a long duration of tourniquet application (from surgical incision to cement setting).

It is hypothesised that tourniquet application during cement fixation only (approximately of 20-30 min duration) will be associated with less pain and impairment than a longer tourniquet application (> 45 minutes).

DETAILED DESCRIPTION:
Background:

Tourniquets are commonly used during total knee replacement (TKR) surgery to provide a bloodless field to improve visualisation [1]. The optimum timing of tourniquet release (ie prior to or after wound closure) has been the subject of many randomised controlled trials with a recent meta-analysis [1] concluding that whilst early release may increase blood loss, it may protect patients from regional complications requiring re-operation such as wound dehiscence, haematomas requiring drainage, knee stiffness and infection. Thus, there is good evidence to suggest that tourniquet use of short duration may be optimal as far as complications are concerned. Few studies have looked at the effect of tourniquet duration on functional recovery, but one [2] observed that quadriceps lag recovered more quickly if short duration tourniquet was used. There has been no research to date on using a tourniquet just during cement fixation of the prosthesis when good visualisation is key to preventing blood-cement mixing. Such an approach is important to investigate as it could further reduce the risks of tourniquet use. However, tourniquet use of such short duration may increase blood loss and increase the risk for donor blood transfusion.

Aim: To establish whether a short duration of tourniquet application (from cement fixation to cement setting)is associated with better outcomes compared to a long duration of tourniquet application (from surgical incision to cement setting).Research Design: A randomised controlled trial will be used to assess the research hypothesis. The research hypothesis is that tourniquet use during cement fixation only will be associated with better physical and functional recovery. However, it may be associated with greater need for donor blood transfusion. Methods: Consenting patients will be randomly allocated to have tourniquet use of either short or long duration in the operating theatre after the patient has been anaesthetised.The tourniquet will be applied at the time of the first skin incision (standard practice for the surgeons involved) for those allocated to the Long-Duration Group, and applied just during cement fixation of the prosthesis for the Short-Duration Group. In both groups, the tourniquet will be removed when the cement has set.

Assessments will be conducted at baseline (up to 6-weeks before surgery during a pre-admission visit), at discharge, then at 2,10, 26 and 52 weeks post surgery. The outcomes of interest include patient-centred measures (Oxford knee score -primary outcome)and other physical measures such as stair climbing test quadriceps lag, and knee range of motion. As the risk of donor blood transfusion may increase with short tourniquet duration, the use of donor blood is also a primary outcome. Reinfusion drains will be used routinely on all patients in order to reduce the need for donor blood. All enrolled patients will undergo a screening leg doppler and another at 2 weeks post surgery for detection of DVTs. Length of stay, and discharge destination (home versus rehabilitation),will also be recorded. Complication type and frequency (including evidence of prosthesis loosening in the first year) will be monitored. The study will be powered to detect a significant difference in Oxford scores. Thus, a sample size of 200 patients will provide sufficient power (80%) at 0.05 significance level to detect a 0.5SD difference in Oxford scores between the 2 treatment arms. This provides for a 20% loss to follow-up and also provides sufficient numbers to detect a large absolute difference (> 20%) in transfusion rate between the groups.

ELIGIBILITY:
Inclusion Criteria:

* primary, unilateral knee replacement;
* capacity to understand the protocol;

Exclusion Criteria:

* inability to read English;
* current warfarin therapy (or similar);
* significant PVD, peripheral arterial disease or diabetes rendering tourniquet use undesirable;
* evidence of chronic or recent DVT in index limb;
* thigh circumference > 100 cm (approximately);
* Jehovah's Witness (ie refusal to receive donor blood)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Oxford Knee score | 10 weeks post surgery
  Oxford knee score is a disease-specific patient perceived knee pain and function survey. It will be collected at baseline (within 2 months of surgery), and then at 10, 26 and 52 weeks post surgery.
Donor blood transfusion rate | Within the acute hospitalisation period (from Day 0 (surgery day), to day of discharge)
  The use of donor blood transfusion in the intra-operative and acute post-operative (hospitalisation) period will be recorded. Criteria for donor blood transfusion is according to the hospital's restrictive transfusion practices.

SECONDARY OUTCOMES:
Knee range of motion (ROM) | ROM will be assessed pre-operatively (within 2 months of surgery), on day 4 post surgery, and at 2, 10,26 and 52 weeks post surgery
  Knee ROM will be assessed photographically according to a method developed by some of the investigators. Photographs taken of the patient's knee in end passive flexion and end passive extension will obtained from the patient in supine. ROM will be measured off the photographs.
Quadriceps lag | Lag will be assessed on Day 4 post surgery, and at 2, 10, 26 and 52 weeks post surgery.
  Quadriceps lag will be assessed with the patient in supine. As for ROM, lag will be measured off photographs. It will be calculated as the difference between full passive knee extension and active extension. Passive end extension will be assessed as previously described. Active extension will be obtained in the same position, but with a towel (or suitable object) under the knee. The patient will attempt to raise their heel off the bed. The knee extension range measured when doing this is called the active extension range.
timed stair test | Measured at 2, 10,26 and 52 weeks post-surgery
  Time (sec)to walk up 10 stairs. Time to walk down 10 stairs. Power will also be calculated from the time together with body weight and step height. The test is not strictly a power test (particularly at 2 weeks)as walking aids/rails can be used as required.
Knee pain | Measured on Day 4 post surgery
  Knee pain measured using a 10cm visual analogue scale
Analgesic consumption | Measured over course of acute care (summation of day 0 to day of discharge)
  The morphine equivalent will be calculated from both PCA and oral analgesic consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Dave, MBBS, Principal Investigator — Surgeon at Fairfield Hospital
Locations (1):
- Fairfield Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Rama KR, Apsingi S, Poovali S, Jetti A. Timing of tourniquet release in knee arthroplasty. Meta-analysis of randomized, controlled trials. J Bone Joint Surg Am. 2007 Apr;89(4):699-705. doi: 10.2106/JBJS.F.00497. PMID 17403789
- [Background] Barwell J, Anderson G, Hassan A, Rawlings I. The effects of early tourniquet release during total knee arthroplasty: a prospective randomized double-blind study. J Bone Joint Surg Br. 1997 Mar;79(2):265-8. doi: 10.1302/0301-620x.79b2.7191. PMID 9119854
- [Derived] Mittal R, Ko V, Adie S, Naylor J, Dave J, Dave C, Harris IA, Hackett D, Ngo D, Dietsch S. Tourniquet application only during cement fixation in total knee arthroplasty: a double-blind, randomized controlled trial. ANZ J Surg. 2012 Jun;82(6):428-33. doi: 10.1111/j.1445-2197.2012.06083.x. Epub 2012 May 10. PMID 22571508